CLINICAL TRIAL: NCT03821532
Title: Evaluation of Adherence and Outcomes in Children With Functional Constipation After Implementing a Constipation Action Plan
Brief Title: Adherence/Outcomes After Use of Constipation Action Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Matthew Di Guglielmo, Clinical Associate Professor of Pediatrics, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 947325
Record Dates: First submitted 2018-12-15; First posted 2019-01-29 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Constipation - Functional
Keywords: Action Plan; Adherence; Pediatrics

STUDY DESIGN:
Intervention Model Description: Control group (standard of care) compared to Intervention group (standard of care plus constipation action plan)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Packet of information containing Standard of Care education materials and {Action Plan or No Action Plan} are prepared prior to enrollment; all participants get unlabeled packet without prior knowledge of participant or investigator or care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Each family will receive a randomized packet containing educational information, rewards charts and an adult literacy test. The treatment plan will be determined based on recommendations from the clinical guidelines for the Evaluation and Treatment of Functional Constipation Infants and Children as published by the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition. At the first visit, the parent(s) will complete an adult literacy test and an initial paper questionnaire regarding symptoms, adherence to the treatment plan and demographics. At 1 month, the primary investigator will call each family and administer a phone survey regarding symptoms and adherence to the treatment plan in the past month. At 3 months, the families will return for a follow up visit with their 3 month reward charts and complete a final paper survey regarding the child's symptoms and adherence to the treatment plan.
- Experimental group (Experimental): Each family will receive a randomized packet containing educational information, rewards charts, an adult literacy test and a constipation action plan tool. The treatment plan will be determined based on recommendations from the clinical guidelines for the Evaluation and Treatment of Functional Constipation Infants and Children as published by the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition. At the first visit, the parent(s) will complete an adult literacy test and an initial paper questionnaire regarding symptoms, adherence to the treatment plan and demographics. At 1 month, the primary investigator will call each family and administer a phone survey regarding symptoms and adherence to the treatment plan in the past month. At 3 months, the families will return for a follow up visit with their 3 month reward charts and complete a final paper survey regarding the child's symptoms, adherence to the treatment plan, and action plan utility.
  Interventions: Other: Constipation Action Plan

INTERVENTIONS:
Other: Constipation Action Plan — Action plan, adapted from Autism Speaks Network, demonstrating Red, Yellow, and Green levels of symptoms with corresponding steps for treatment or action by parent/guardian, tailored by care provider to the child's condition.
  Arms: Experimental group

SUMMARY:
Adherence to recommendations for treatment of chronic constipation in pediatric population is often poor. This study is attempting to improve adherence, and outcomes, by implementing a trial of a constipation action plan plus standard of care, compared to standard of care alone, in an outpatient pediatric population.

DETAILED DESCRIPTION:
Functional Constipation is a common childhood problem. The goal of this study is to evaluate if a constipation action plan had any impact on improved adherence in management. Children are eligible to participate in the study if they are otherwise healthy children whose primary language is English with no conditions that would predispose them to develop constipation, between the ages of 3 and 8 years of age and if they meet the ROME IV criteria for functional constipation. The primary objective is to assess compliance in pediatric patients with functional constipation that have been provided a constipation action plan plus educational information. The secondary objectives are to assess improvement of constipation symptoms in pediatric patients with functional constipation that have been provided a constipation action plan and educational information and to assess the perceived effectiveness of the constipation action plan from the viewpoint of the family. The proposed study hypothesizes that patients diagnosed with functional constipation will have improved adherence to medication treatment plan, to fiber intake, and to toilet sit time and have improved constipation symptoms overall when provided with both a constipation action plan and educational information regarding dietary changes, toilet sit time, and medications as compared to education information alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* History of functional constipation
* English as primary language

Exclusion Criteria:

* History of medical conditions pre-disposing to constipation
* English as a second language
* Chronic gastrointestinal disease

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Compliance Questionnaire | At screening
  Evaluate compliance using the constipation/adherence questionnaire. The questionnaire has 3 questions addressing the total number of days missed per week taking the prescribed medications, toilet sit times and dietary intake
Compliance Questionnaire | 1 Month
  Compliance will be evaluated by reviewing the sticker reward chart at the 3 month visit and calculating the number of days the child missed medication dose, did not sit on the toilet as instructed and how many days were missed of adequate fiber intake. Further evaluate compliance using the constipation/adherence questionnaire. The questionnaire has 3 questions addressing the total number of days missed per week taking the prescribed medications, toilet sit times and dietary intake
Compliance Questionnaire | 3 Month
  Compliance will be evaluated by reviewing the sticker reward chart at the 3 month visit and calculating the number of days the child missed medication dose, did not sit on the toilet as instructed and how many days were missed of adequate fiber intake. Further evaluate compliance using the constipation/adherence questionnaire. The questionnaire has 3 questions addressing the total number of days missed per week taking the prescribed medications, toilet sit times and dietary intake
Compliance Reward Chart | 3 Month
  Compliance will be evaluated by reviewing the sticker reward chart at the 3 month visit and calculating the number of days the child missed medication dose, did not sit on the toilet as instructed and how many days were missed of adequate fiber intake.

SECONDARY OUTCOMES:
Symptoms | At screening
  Number of participants with positive constipation symptoms using ROME IV Criteria
Symptoms | 1 Month
  Number of participants with positive constipation symptoms using ROME IV Criteria
Symptoms | 3 Month
  Number of participants with positive constipation symptoms using ROME IV Criteria
Perceived effectiveness | 1 month telephone encounter
  Anonymous survey addresses questions regarding the number of days the child was in each zone of the constipation action plan and whether or not the plan helped the family better manage the child's symptoms, decreased calls to the physician and whether or not it was easy to use.
Perceived effectiveness | 3 month follow up visit
  Anonymous survey addresses questions regarding the number of days the child was in each zone of the constipation action plan and whether or not the plan helped the family better manage the child's symptoms, decreased calls to the physician and whether or not it was easy to use.
Caregiver Literacy | 0 months
  Assess literacy level for caregivers by administering the Short-Form Rapid Assessment of Adult Literacy in Medicine. Final score of 0, 1-3, 4-6, or 7 determines grade reading level (3rd grade or less, 4th to 6th, 7th to 8th, 9th grade and higher). There is no better or worse outcome, just stratification of literacy (medical) is determined.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Di Guglielmo, MD PhD, Principal Investigator — Nemours
Locations (1):
- Alfred I. duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palsson OS, Whitehead WE, van Tilburg MA, Chang L, Chey W, Crowell MD, Keefer L, Lembo AJ, Parkman HP, Rao SS, Sperber A, Spiegel B, Tack J, Vanner S, Walker LS, Whorwell P, Yang Y. Rome IV Diagnostic Questionnaires and Tables for Investigators and Clinicians. Gastroenterology. 2016 Feb 13:S0016-5085(16)00180-3. doi: 10.1053/j.gastro.2016.02.014. Online ahead of print. PMID 27144634
- [Background] van den Berg MM, Benninga MA, Di Lorenzo C. Epidemiology of childhood constipation: a systematic review. Am J Gastroenterol. 2006 Oct;101(10):2401-9. doi: 10.1111/j.1572-0241.2006.00771.x. PMID 17032205
- [Background] Steiner SA, Torres MR, Penna FJ, Gazzinelli BF, Corradi CG, Costa AS, Ribeiro IG, de Andrade EG, do Carmo Barros de Melo M. Chronic functional constipation in children: adherence and factors associated with drug treatment. J Pediatr Gastroenterol Nutr. 2014 May;58(5):598-602. doi: 10.1097/MPG.0000000000000255. PMID 24345842
- [Background] Graves MM, Roberts MC, Rapoff M, Boyer A. The efficacy of adherence interventions for chronically ill children: a meta-analytic review. J Pediatr Psychol. 2010 May;35(4):368-82. doi: 10.1093/jpepsy/jsp072. Epub 2009 Aug 26. PMID 19710248
- [Background] Luersen K, Davis SA, Kaplan SG, Abel TD, Winchester WW, Feldman SR. Sticker charts: a method for improving adherence to treatment of chronic diseases in children. Pediatr Dermatol. 2012 Jul-Aug;29(4):403-8. doi: 10.1111/j.1525-1470.2012.01741.x. Epub 2012 Apr 4. PMID 22471987
- [Background] Ismail N, Ratchford I, Proudfoot C, Gibbs J. Impact of a nurse-led clinic for chronic constipation in children. J Child Health Care. 2011 Sep;15(3):221-9. doi: 10.1177/1367493511406568. Epub 2011 Aug 9. PMID 21828166
- [Background] Arozullah AM, Yarnold PR, Bennett CL, Soltysik RC, Wolf MS, Ferreira RM, Lee SY, Costello S, Shakir A, Denwood C, Bryant FB, Davis T. Development and validation of a short-form, rapid estimate of adult literacy in medicine. Med Care. 2007 Nov;45(11):1026-33. doi: 10.1097/MLR.0b013e3180616c1b. PMID 18049342

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03821532/Prot_SAP_000.pdf